CLINICAL TRIAL: NCT06491160
Title: A Trial to Explore Performance and FMRI BOLD Signal Changes During Impulsivity Tasks in Impulsive Patients with Attention Deficit Hyperactivity Disorder and Borderline Personality Disorder
Brief Title: Performance and FMRI BOLD Signal Changes in Impulsive Patients
Status: Completed | Type: Observational
Sponsor: Simone Grimm (Other)
Collaborators: Charité Research Organisation GmbH (Other); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Simone Grimm, Prof. Dr. habil., Medical School Berlin
Organization: Medical School Berlin (Other)
Other Study IDs: MSBC004
Record Dates: First submitted 2024-06-06; First posted 2024-07-08 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; Borderline Personality Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Borderline Personality Disorder; Functional Brain Changes; BOLD responses
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Attention Deficit Hyperactivity Disorder: Subjects eligible for enrolment in this study must the following criteria:
  1. meet current Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for ADHD as a primary diagnosis as assessed by the Structured Clinical Interview for DSM Disorders (SCID) and the Structured Clinical Interview for DSM Personality Disorders (SCID-PD)
  2. between 18 and 45 years, inclusive
  3. BIS-11 score of ≥ 70
- Borderline Personality Disorder: Subjects eligible for enrolment in this study must meet all of the following criteria:
  1. meet current DSM-5 criteria for BPD as a primary diagnosis as assessed by SCID and SCID-PD
  2. between 18 and 45 years, inclusive
  3. BIS-11 score of ≥ 70

SUMMARY:
This study is a preceding study conducted to validate the methodology for assessing impulsivity by tasks and task-based fMRI measurements in patients with Attention Deficit Hyperactivity Disorder (ADHD) or Borderline Personality Disorder (BPD).

DETAILED DESCRIPTION:
It is planned to conduct a clinical trial to test pharmacodynamic effects of a new drug under development for impulsivity including patients with ADHD or BPD. For the preparation of this planned trial, a preceding study will be conducted. The results of this preceding study will be needed to prepare and plan the upcoming proof-of-clinical-principle-study regarding behavioral effects, involved brain regions, effect sizes, patient experience, and task design. Testing and optimizing the study procedures in advance in this preceding study will help to define the objectives and endpoints of the planned pharmacodynamic trial.

ELIGIBILITY:
Inclusion Criteria:

1. meet current DSM-5 criteria for ADHD or BPD as a primary diagnosis as assessed by SCID and SCID-PD
2. between 18 and 45 years, inclusive
3. BIS-11 score of ≥ 70
4. completely fluent German speaker who, in the opinion of the Investigator, is capable of completing the fMRI and behavioral tasks
5. must have signed the informed consent form prior to the first study-related procedure indicating they understand the purpose of, and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Lifetime diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I or II disorder, delusional disorder, or autism spectrum disorder as confirmed by the SCID at screening visit
2. Moderate or severe substance use disorder within the last 6 months.
3. Any other psychiatric disorder that is not currently stable in symptoms and treatment. Stable is defined as have no significant changes in symptom acuity or medication treatment in the 3 months prior to enrollment
4. Positive results on a urine drug screen or alcohol breath test, or any signs or symptoms of acute intoxication at screening or enrollment visit
5. A female subject with a positive pregnancy test at screening or enrollment visit
6. Unstable medical condition, history of seizure disorders, stroke, brain tumor, or any other major neurological illness
7. Subjects deemed to be at significant risk of serious violence or suicide based on any one of the following:

   * Significant risk of committing violent acts, homicide, serious self-harm, or suicide based on history, routine psychiatric status examination, or according to the investigator's experience OR
   * Any suicide attempt in the past 6 months (i.e. actual attempt, interrupted attempt, aborted attempt) prior to enrollment OR
   * Any suicidal ideation of type 4 or 5 in the Columbia-Suicide Severity Rating Scale (C-SSRS) in the past 6 months prior to enrollment
8. Subjects not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (that, in the investigator's opinion, makes the subject an unreliable trial subject)
9. Concomitant use of restricted psychotropic medication. All restricted psychotropic medications must be washed out at least 5 half-lives prior to enrollment (including ADHD medications such as amphetamine or methylphenidate derivates). Allowed medications must be stable in agent, dose, and frequency for > 3 month prior to enrollment:

   * a single antidepressant of the Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin-Noradrenaline Reuptake Inhibitor (SNRI) class
   * A single second-generation antipsychotic at a low dose (1 thorazine dose equivalent or less, which translates to ≤ 2 mg/day for risperidone, 5 mg/day for olanzapine, 75 mg/day for quetiapine, 60 mg/day for ziprasidone, and 7.5 mg/day for aripiprazole)
   * Permitted sleep medications must be nightly scheduled medications (not PRN) and may include non-benzodiazepines, antihistamines, melatonin, trazodone, low dose doxepin (≤ 50mg), and low dose quetiapine (≤75mg qhs).
10. Any contraindication to undergo an MRI radiography (e.g. history of surgery involving metal implants), including but not limited the following:

    * A planned medical treatment within the study period that might interfere with the study procedures
    * Subjects who have undergone operations to the head
    * Subjects with significant hearing impairments which, in the opinion of the investigator, may interfere with the performance of fMRI tasks
    * Subjects with a significant visual impairment including color blindness, or history of ocular treatment including corrective laser eye surgery, or ongoing condition, which in the opinion of the investigator may interfere with the performance of the behavioral or fMRI tasks
11. Subject is a staff member or the relative of a staff member or is in a subordinate relationship with the Investigator
12. Signs or symptoms of Post-Covid disease
13. Inability or unwillingness to comply with study procedures, including study prohibitions and restrictions
14. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
15. Vulnerable subject who lives in an institution on court or authority order
16. Participation in another clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population includes individuals diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) and with Borderline Personality Disorder (BPD). Subjects must meet current DSM-5 criteria for ADHD or BPD as a primary diagnosis as assessed by SCID and SCID-PD. Subjects must score higher than 70 on the Barratt Impulsiveness Scale (BIS) to be included in the study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Average percent BOLD signal change during the 4-Choice Serial-Reaction Time Task (4-CSRTT) | During the 4-CSRTT on experimental day (visit number 2 (study day 1))
  Blood oxygen level dependent (BOLD) fMRI signal changes will be analyzed to identify brain regions with significant activation during the 4-CSRTT
Average percent BOLD signal change during the Stop Signal Task (SST) | During the SST on experimental day (visit number 2 (study day 1))
  Blood oxygen level dependent (BOLD) fMRI signal changes will be analyzed to identify brain regions with significant activation during the SST
Average percent BOLD signal change during resting state | During resting state on experimental day (visit number 2 (study day 1))
  Blood oxygen level dependent (BOLD) fMRI signal magnitude and BOLD signal standard deviation during resting state
Assessment of brain perfusion | During asl on experimental day (visit number 2 (study day 1))
  Change in relative and absolute cerebral blood flow are measured through Arterial Spin Labeling (ASL)

OTHER OUTCOMES:
Correlation between BOLD signal during the 4-CSRTT and impulsivity scores on the BIS-11 | Impulsivity scores were assessed on the screening day (visit number 1 (study days -28 to -1)), while BOLD signal changes during the 4-CSRTT were measured on the experimental day (visit number 2 (study day 1))
  Correlation between magnitude of BOLD signal during the 4-CSRTT and impulsivity scores on the BIS-11
Correlation between BOLD signal during the SST and impulsivity scores on the BIS-11 | Impulsivity scores were assessed on the screening day (visit number 1 (study days -28 to -1)), while BOLD signal changes during the SST were measured on the experimental day (visit number 2 (study day 1))
  Correlation between magnitude of BOLD signal during the SST and impulsivity scores on the BIS-11
Correlation between BOLD signal during the 4-CSRTT and impulsivity scores on the S-UPPS | Impulsivity scores were assessed on the screening day (visit number 1 (study days -28 to -1)), while BOLD signal changes during the 4-CSRTT were measured on the experimental day (visit number 2 (study day 1))
  Correlation between magnitude of BOLD signal during the 4-CSRTT and impulsivity scores on the S-UPPS
Correlation between BOLD signal during the SST and impulsivity scores on the S-UPPS | Impulsivity scores were assessed on the screening day (visit number 1 (study days -28 to -1)), while BOLD signal changes during the SST were measured on the experimental day (visit number 2 (study day 1))
  Correlation between magnitude of BOLD signal during the SST and impulsivity scores on the S-UPPS
Reaction times in ms | During all tasks on experimental day (visit number 2 (study day 1))
  Reaction times in ms extracted from the in- scanner protocol log files
Premature responses | During all tasks on experimental day (visit number 2 (study day 1))
  Number of premature responses extracted from the in- scanner protocol log files
Reaction times during the 4-CSRTT after stress induction | During the 4-CSRTT after stress is induced on experimental day (visit number 2 (study day 1))
  Task performance is measured based on the reaction times (RTs) for choices. Stress is induced using the Mannheim Multicomponent Stress Test (MMST).
Premature responses during the 4-CSRTT after stress induction | During the 4-CSRTT after stress is induced on experimental day (visit number 2 (study day 1))
  Task performance is measured based on the number of premature responses. Stress is induced using the Mannheim Multicomponent Stress Test (MMST).
Impulsive choice ratio during the 4-CSRTT after stress induction | During the 4-CSRTT after stress is induced on experimental day (visit number 2 (study day 1))
  Task performance is measured based on the impulsive choice ratio. Stress is induced using the Mannheim Multicomponent Stress Test (MMST).
Reaction times during the DDT after stress induction | During the DDT after stress is induced on experimental day (visit number 2 (study day 1))
  Task performance is measured based on reaction times (RTs) for choices. Stress is induced using the Mannheim Multicomponent Stress Test (MMST).
Premature responses during the DDT after stress induction | During the DDT after stress is induced on experimental day (visit number 2 (study day 1))
  Task performance is measured based on the number of premature responses. Stress is induced using the Mannheim Multicomponent Stress Test (MMST).
Correlation between BOLD signal and behavioral measures during 4-CSRTT | during the 4-CSRTT conducted in the scanner on experimental day (visit number 2 (study day 1))
  Correlation between magnitude of BOLD signal during 4-CSRTT and behavioral measures of the 4-CSRTT
Correlation between BOLD signal and behavioral measures during SST | during the SST conducted in the scanner on experimental day (visit number 2 (study day 1))
  Correlation between magnitude of BOLD signal during SST and behavioral measures of the SST

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keicher, Dr. med., Principal Investigator — Charité Research Organisation, Berlin, Germany
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No